CLINICAL TRIAL: NCT07120698
Title: Adaptive Adjuvant Sintilimab Therapy Guided by MRD in II-IIIB Stage NSCLC Patients With Non-pCR Pathological Response After Neoadjuvant Immunotherapy Combined With Chemotherapy: a Prospective, Multi-center, Single-arm, Phase II Trial
Brief Title: Adaptive Adjuvant Sintilimab Therapy Guided by MRD (ADAPT Lung)
Acronym: CTONG 2508
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Association of Clinical Trials (Other)
Collaborators: Zunyi Medical College (Other); Suining Central Hospital (Other); Shenzhen Second People's Hospital (Other); Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Yi Yang, chief physician, Guangdong Association of Clinical Trials
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-S-174
Record Dates: First submitted 2025-07-08; First posted 2025-08-13 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: NSCLC (Non-small Cell Lung Cancer); MRD; II-IIIB Stages; Adjuvant Immunotherapy
Keywords: MRD; II-IIIB stages; NSCLC (non-small cell lung cancer); adjuvant immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sintilimab

STUDY DESIGN:
Intervention Model Description: Model Description
Masking Description: Masking Description
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): sintilimab
  Interventions: Drug: Sintilimab

INTERVENTIONS:
Drug: Sintilimab — Patients who met the inclusion criteria were treated with adaptive adjuvant sintilimab therapy guided by MRD.
  Patients should test twice at postoperative days 3 to 7 and again at postoperative day 28 (±3 days). The results of these two tests will be used to determine the subsequent treatment pathway. Participants with two consecutive positive MRD tests or a single positive MRD test will be enrolled in the MRD+ treatment cycle：they will receive adjuvant treatment with sintilimab (200 mg, intravenous infusion, every 3 weeks). Follow-up visits will be conducted every 3 months, during which chest CT scans and MRD testing will be performed. If MRD becomes negative, treatment will be discontinued and the participant will be monitored. If MRD remains positive, treatment with sintilimab will continue.
  Participants with two consecutive negative MRD tests will be enrolled in the MRD- treatment cycle：they will undergo follow-up observation only. Follow-up visits will be conducted every 3 months

SUMMARY:
This is a multicenter, prospective, open-label Phase II study designed to evaluate the safety and efficacy of adjuvant sintilimab therapy guided by minimal residual disease (MRD) in patients with Stage II-IIIB non-small cell lung cancer (NSCLC) who have not achieved a pathological complete response (non-pCR) after neoadjuvant immunotherapy combined with chemotherapy. The study is being conducted at the Third People's Hospital of Chengdu and the Guangdong Provincial People's Hospital.

DETAILED DESCRIPTION:
Patients with Stage II-IIIB NSCLC who have not achieved a pathological complete response after neoadjuvant immunotherapy combined with chemotherapy will be enrolled in this study. Eligible patients will receive adjuvant sintilimab therapy guided by MRD.

Patients should undergo a test 3 to 7 days after surgery, and another test 28 days (±3 days) after. surgery The results of these two tests will be used to determine the subsequent treatment pathway. Participants with two consecutive positive MRD test results or a single positive MRD test result will be included in the MRD + treatment cycle: they will receive adjuvant therapy with sintilimab (200 mg, intravenous infusion, every 3 weeks). Follow-up will be conducted every 3 months, during which chest CT scans and MRD tests will be performed. If the MRD test result turns negative, treatment will be discontinued and participants will be monitored. If the MRD test result remains positive, sintilimab treatment will continue.

Participants with two consecutive negative MRD test results will be included in the MRD - treatment cycle: they will only receive follow-up observation. Follow-up will be conducted every 3 months, during which chest CT scans and MRD tests will be performed. If the MRD test result turns positive, adjuvant therapy with sintilimab (200 mg, intravenous infusion, every 3 weeks) will be initiated. If the MRD test result remains negative, follow-up observation will continue.

The maximum number of treatment cycles for sintilimab therapy is 18 cycles. Safety will be evaluated through adverse events (AE) and laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent prior to the initiation of any trial-related procedures.
2. Male or female aged ≥18 years and ≤75 years.
3. Histologically or cytologically confirmed non-small cell lung cancer (NSCLC).
4. Received 3-4 cycles of neoadjuvant immunotherapy (PD-1 inhibitor) combined with chemotherapy.
5. Underwent radical surgical treatment (R0), with surgical procedures including lobectomy or sleeve lobectomy. All gross tumors must be completely resected at the end of surgery, and all surgical margins of the resected tumors must be negative. Systemic lymph node dissection is required.
6. Clinical stage II, IIIA, or IIIB (limited to resectable N2) according to the AJCC 8th edition TNM classification for lung cancer. Resectable N2 refers to non-massive (defined as short-axis diameter <3 cm), discrete, or single-station N2 involvement. If clinically suspected of N2 or N3, pathological confirmation is recommended whenever feasible.
7. Patients with pathological response assessment of 1%-90% residual viable tumor (RVT).
8. No EGFR mutations, ROS1 fusions, ALK fusions, or RET fusions. Other potentially targetable driver gene alterations will be determined in consultation with the sponsor.
9. No prior anti-tumor treatment other than PD-1 inhibitors and chemotherapy before radical surgery for lung cancer.
10. Completed radical surgery for lung cancer 4-12 weeks prior to study enrollment, with pathological confirmation of R0 resection and radiological evidence of no residual tumor foci 1 month after radical surgery.
11. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
12. Life expectancy >6 months.
13. Adequate organ function:

1. Absolute neutrophil count (ANC) ≥1.5×10^9/L without the use of granulocyte colony-stimulating factor within the past 14 days.

2. Platelets ≥100×10^9/L without transfusion within the past 14 days. 3. Hemoglobin >9 g/dL without transfusion or use of erythropoiesis-stimulating agents within the past 14 days.

4. Total bilirubin ≤1.5× upper limit of normal (ULN). 5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN (subjects with liver metastases are allowed to have ALT or AST ≤5×ULN).

6. Serum creatinine ≤1.5×ULN and creatinine clearance (calculated using the Cockcroft-Gault formula) ≥60 ml/min.

7. Good coagulation function, defined as international normalized ratio (INR) or prothrombin time (PT) ≤1.5×ULN.

8. Normal thyroid function, defined as thyroid-stimulating hormone (TSH) within the normal range. Subjects with baseline TSH outside the normal range are eligible if total T3 (or free T3) and free T4 are within the normal range.

9. Cardiac enzyme profile within the normal range (subjects with isolated laboratory abnormalities deemed not clinically significant by the investigator are also eligible).

14. For female subjects of childbearing potential, a negative urine or serum pregnancy test must be obtained within 3 days prior to the first administration of the study drug (Day 1 of Cycle 1). If the urine pregnancy test result is inconclusive, a serum pregnancy test is required. Postmenopausal women are defined as those who have been amenorrheic for at least 1 year, or those who have undergone surgical sterilization or hysterectomy.

15. All subjects (regardless of gender) at risk of conception must use contraception with a failure rate of less than 1% per year throughout the treatment period until 120 days after the last administration of the study drug (or 180 days after the last administration of chemotherapy).

16. Provide samples for MRD assessment (surgical tissue + blood).

Exclusion Criteria:

1. Diagnosis of any malignancy other than non-small cell lung cancer within 5 years prior to the first dose (excluding completely treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or carcinoma in situ that has been completely resected).
2. Received adjuvant radiotherapy prior to dosing.
3. Patients who underwent pneumonectomy.
4. Currently participating in an interventional clinical study or received other investigational drugs or used investigational devices within 4 weeks prior to the first dose.
5. Received neoadjuvant treatment with anti-tumor therapies other than chemotherapy and immunotherapy.
6. Presence of unhealed surgical incisions, ulcers, or fractures.
7. In the investigator's opinion, severe concomitant systemic diseases that may affect the subject's ability to complete the study. Subjects with positive autoimmune antibodies must be assessed and confirmed by the investigator to have no autoimmune diseases requiring systemic treatment before enrollment.
8. Presence of primary immunodeficiency diseases.
9. Receiving systemic corticosteroid therapy within 7 days prior to the first dose of the study (excluding intranasal, inhaled, or other topical corticosteroids). Note: The use of physiologic doses of corticosteroids (≤10 mg/day prednisone or equivalent) is permitted.
10. Known allogeneic organ transplantation (excluding corneal transplantation) or allogeneic hematopoietic stem cell transplantation.
11. Known allergy to the active ingredient or excipients of the study drug, sintilimab.
12. Not fully recovered from toxicities and/or complications caused by any prior interventions prior to the start of treatment (i.e., ≤Grade 1 or returned to baseline, excluding fatigue or alopecia).

Ages: 28 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2029-06-26 (Estimated); Study Completion 2029-07-26 (Estimated)

PRIMARY OUTCOMES:
2-year EFS rate | 2 year after treatment initiation
  Event-free survival (EFS) is defined as the time from the date of randomization (or the start of treatment) to the first occurrence of any of the following events: disease progression, local or distant recurrence, or death due to any cause. If a patient does not experience any of these events within 2 years, they are considered to have achieved 2-year EFS.

SECONDARY OUTCOMES:
mEFS | From enrollment to disease progression, reoccurrence, or death due to any cause. (Up to a median of 30 months)
  The median Event-Free Survival (mEFS) is defined as the median time from the date of randomization or the initiation of treatment to the first occurrence of a prespecified event, such as disease progression, death, or change in treatment regimen.
2-year OS rate | 24 months
  The 2-year Overall Survival (OS) rate is defined as the proportion of patients who remain alive at the specific time point of 2 years from the date of randomization or the initiation of treatment.
mOS | OS is defined as the time from enrollment to death, regardless of disease recurrence, assessed up to 100 months
  The median overall survival (mOS) is defined as from date of enrollment until the date of first documented date of death from any cause, whichever came first, assessed up to 40 months, at which the survival rate is 50%.
AEs | 24 months
  Safety and tolerability will be assessed by the incidence of adverse events (AEs), serious adverse events (SAEs), immune-related adverse events (irAEs), deaths, and laboratory abnormalities.
QoL | 24 months
  Per physician's discretion, the patient will complete one or more of the following QoL instruments:
  EQ-5D is a 5 item questionnaire with a total score ranging from 0 to 100 with the higher score indicating greater satisfaction, EORTC QLQ-C30 is a 30 item questionnaire with a total score ranging from 1 to 4 with the lower score indicating greater satisfaction.

OTHER OUTCOMES:
Analyze the proportion of the four types of pathological response (1%-5% irRVT vs. >5%-30% irRVT vs. >30%-80% irRVT vs. >80% irRVT) and their correlation with median event-free survival (mEFS). | From enrollment to disease progression, reoccurrence, or death due to any cause. (Up to a median of 30 months)
  Proportion of the four types of RVT results Assessment of the relationship between different RVT results and median event-free survival (mEFS)

CONTACTS AND LOCATIONS:
Overall Officials: Yang, Principal Investigator — Guangdong Association of Clinical Trials
Locations (2):
- China (2):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The third people's hospital of chengdu, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No
We will not share individual participant data (IPD) because the original informed-consent forms signed by participants did not explicitly cover secondary use of their data by external parties, and thus sharing IPD would risk violating the approved ethics agreement.